CLINICAL TRIAL: NCT03537664
Title: Analysis of Metabolically Active Bacteria After Adjunctive Steps for Disinfection of Teeth With Primary Endodontic Infections: RNA- and DNA-based Molecular Study
Brief Title: Adjunctive Steps for Disinfection of Teeth With Primary Endodontic Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ericka Tavares Pinheiro, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2016/15473-0
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Periapical Periodontitis; Bacterial Infections
Keywords: Periapical Periodontitis; Bacterial Infections; Root Canal Preparation; Calcium Hydroxide; Real-Time Polymerase Chain Reaction; RNA-Directed DNA Polymerase
MeSH Terms: conditions — Periapical Periodontitis; Bacterial Infections | interventions — Root Canal Preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total bacteria analysis after 1rst- and 2nd-visit procedures (Experimental): DNA levels and activity (RNA/DNA ratio) of total bacteria after the first-visit procedures (root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation) and the second-visit protocol (intracanal medication with calcium hydroxide paste, followed by an 2nd-visit root canal preparation). Additionally, the composition of the active microbiome will be assessed by Next Generation Sequencing (NGS) analysis of the root canal samples, and the success rate (apical repair) of the endodontic treatment after 1 follow-up period will be assessed by an intraoral radiograph and cone beam computed tomography (CBCT) analyses.
  Interventions: Procedure: Root canal preparation; Procedure: Intracanal medication
- Bacterial species analysis after root canal preparation (Other): DNA levels and activity (RNA/DNA ratio) of Bacteroidaceae sp. 272 , Cutibacterium acnes, Selenomonas spp., and Enterococcus faecalis after root canal preparation.Additionally, the success rate (apical repair) of the endodontic treatment after 1 follow-up period will be assessed by an intraoral radiograph and cone beam computed tomography (CBCT) analyses.
  Interventions: Procedure: Root canal preparation

INTERVENTIONS:
Procedure: Root canal preparation — First endodontic treatment session includes the root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation.
Procedure: Intracanal medication — The second endodontic treatment includes the intracanal medication with calcium hydroxide paste, followed by an 2nd-visit root canal preparation
  Arms: Total bacteria analysis after 1rst- and 2nd-visit procedures

SUMMARY:
This study aims to evaluate an endodontic treatment protocol using adjunctive steps for disinfection of teeth with primary endodontic infections.

DETAILED DESCRIPTION:
The success of endodontic treatment in teeth with necrotic pulp and apical periodontitis depends on the reduction of viable microorganisms of root canals by endodontic disinfection procedures. This study aims to evaluate by molecular methods the effect of different disinfection procedures on reduction, diversity and microbial metabolic activity. Patients with necrotic pulps and apical periodontitis in single-rooted teeth will be selected. Microbiological samples will be taken from root canals after access cavity (S1), after chemomechanical preparation with Reciproc System and 2.5% NaOCl (S2), after irrigant activation using the XP-Endo Finisher instrument (S3a) and ultrasonic activation (S3b); and after intracanal medication with calcium hydroxide for 14 days (S4), followed by 2nd-visit root canal preparation (S5). DNA and RNA will be extracted from root canal samples, and complementary DNA (cDNA) synthetized using reverse transcription reaction. The effect of treatment protocols on total microbiota levels will be determined by DNA-based quantitative polymerase chain reaction (qPCR) using universal primers for Bacteria domain. RNA of root canal samples will be used to determine the diversity of metabolically active microbiota by Reverse Transcriptase Reaction (RT), followed by amplification (PCR) and high throughput sequencing of the hypervariable region V4-V5 of 16S rRNA gene. The metabolic activity of the most prevalent species / taxa will be calculated by rRNA- and DNA-based molecular methods. Ratios between rRNA and DNA levels will be calculated to search for active bacteria (rRNA/DNA ≥ 1) in root canal samples. Data will be analyzed by statistical tests, with 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with necrotic pulps and asymptomatic apical periodontitis

Exclusion Criteria:

* patients who had received antibiotics during the previous 3 months or had any general disease,
* teeth that could not be properly isolated with rubber dam,
* non-restored teeth,
* periodontal pockets depths greater than 4 mm,
* previous endodontic treatment,
* open apex,
* crown/root fracture
* root resorption or calcifications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ericka T Pinheiro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Samples from 20 patients were used for the analysis of total bacteria in 1st and 2nd visits. Additional 25 patients were necessary for the analysis of specific bacterial species in post-instrumentation samples (n=45 patients).
Groups:
- Bacterial Species Analysis After Root Canal Preparation: DNA levels and activity (RNA/DNA ratio) of Bacteroidaceae sp. 272 , Cutibacterium acnes, Selenomonas spp., and Enterococcus faecalis after root canal preparation. Additionally, the success rate (apical repair) of the endodontic treatment after 1 follow-up period will be assessed by an intraoral radiograph and cone beam computed tomography (CBCT) analyses.
Period: Overall Study
Arm/Group | Total Bacteria Analysis After 1rst- and 2nd-visit Procedures | Bacterial Species Analysis After Root Canal Preparation
Started | 20 | 25
Metabolic Activity of Bacteria | 15 (5 patients were excluded from metabolic activity analysis (lost of RNA)) | 25
Bacterial Levels | 20 | 25
Bacterial Community Diversity | 10 | 0
Endodontic Success | 20 | 10
Completed | 20 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Root Canal Preparation and Medication: First endodontic treatment session includes the root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation. The second endodontic treatment includes the intracanal medication with calcium hydroxide paste.
  Root canal preparation: First endodontic treatment session includes the root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation.
  Intracanal medication: The second endodontic treatment includes the intracanal medication with calcium hydroxide paste.
Arm/Group | Root Canal Preparation and Medication
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 41 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 45
Region of Enrollment [Number; unit: participants]
  Brazil | 45
Number of participants with infected root canals [Count of Participants; unit: Participants] | 45

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Activity of Persistent Bacteria
Description: The metabolic activity (rRNA/DNA ratio) of total bacteria, Bacteroidaceae sp. 272, Cutibacterium acnes, Selenomonas spp. and Enterococcus faecalis in root canal samples taken before and after endodontic procedures.
Time Frame: After 14 day treatment period
Population: There was a lost of RNA samples from 5 cases.
Measure: Mean (Standard Deviation); unit: RNA/DNA ratio
Groups:
- Total Bacteria Analysis After 1rst- and 2nd-visit Procedures: RNA/DNA ratio of total bacteria after the first- and second-visit treatment (active bacteria with rRNA/DNA ≥ 1). First endodontic treatment session includes the root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation. The second endodontic treatment includes the intracanal medication with calcium hydroxide paste for 14 days, followed by an 2nd-visit root canal preparation.
- Bacterial Species Analysis After Root Canal Preparation: RNA/DNA ratio of Bacteroidaceae sp. 272 , Cutibacterium acnes, Selenomonas spp., and Enterococcus faecalis after root canal preparation (active bacteria with rRNA/DNA ≥ 1).
Arm/Group | Total Bacteria Analysis After 1rst- and 2nd-visit Procedures | Bacterial Species Analysis After Root Canal Preparation
Number analyzed (Participants) | 15 | 20
RNA/DNA ratio
  Total bacteria at baseline (S1): number analyzed (Participants) | 15 | 0
  Total bacteria at baseline (S1) | 4.748 (6.2904) |
  Total bacteria after root canal Preparation (S2): number analyzed (Participants) | 15 | 0
  Total bacteria after root canal Preparation (S2) | 2.57 (3.21) |
  Total bacteria after adjunctive procedures (S3): number analyzed (Participants) | 15 | 0
  Total bacteria after adjunctive procedures (S3) | 2.614 (2.978) |
  Total bacteria after intracanal medication (S4): number analyzed (Participants) | 15 | 0
  Total bacteria after intracanal medication (S4) | 4.0008 (4.374) |
  Total bacteria after 2nd-visit preparation (S5): number analyzed (Participants) | 15 | 0
  Total bacteria after 2nd-visit preparation (S5) | 3.7875 (2.9727) |
  Bacteroidaceae sp. HOT-272 at S1: number analyzed (Participants) | 0 | 20
  Bacteroidaceae sp. HOT-272 at S1 |  | 1.136 (0.1318)
  Bacteroidaceae sp. HOT-272 at S2: number analyzed (Participants) | 0 | 20
  Bacteroidaceae sp. HOT-272 at S2 |  | 1.123 (0.1033)
  Cutibacterium acnes at S1: number analyzed (Participants) | 0 | 20
  Cutibacterium acnes at S1 |  | 1.411 (0.3693)
  Cutibacterium acnes at S2: number analyzed (Participants) | 0 | 20
  Cutibacterium acnes at S2 |  | 1.489 (0.3547)
  Selenomonas spp. at S1: number analyzed (Participants) | 0 | 20
  Selenomonas spp. at S1 |  | 1.092 (0.09859)
  Selenomonas spp. at S2: number analyzed (Participants) | 0 | 20
  Selenomonas spp. at S2 |  | 1 (0)
  Enterococcus faecalis at S1: number analyzed (Participants) | 0 | 20
  Enterococcus faecalis at S1 |  | 0.7433 (0.1882)
  Enterococcus faecalis at S2: number analyzed (Participants) | 0 | 20
  Enterococcus faecalis at S2 |  | 0 (0)

2. Secondary Outcome: Bacterial Levels
Description: Quantitative data of total bacteria, Bacteroidaceae sp. HOT-272, Cutibacterium acnes, Selenomonas spp. and Enterococcus faecalis determined by DNA-based qPCR (quantitative polymerase chain reaction).
Time Frame: After 14 day treatment period
Population: There was a lost of RNA samples from 5 cases
Measure: Median (Full Range); unit: DNA copies (Bacterial levels)
Groups:
- Total Bacteria Analysis After 1rst- and 2nd-visit Procedures: DNA levels of total bacteria after the first-visit procedures (root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation) and the second-visit protocol (intracanal medication with calcium hydroxide paste, followed by an 2nd-visit root canal preparation).
- Bacterial Species Analysis After Root Canal Preparation: DNA levels of Bacteroidaceae sp. 272 , Cutibacterium acnes, Selenomonas spp., and Enterococcus faecalis after root canal preparation.
Arm/Group | Total Bacteria Analysis After 1rst- and 2nd-visit Procedures | Bacterial Species Analysis After Root Canal Preparation
Number analyzed (Participants) | 20 | 20
DNA copies (Bacterial levels)
  Total bacteria at baseline (S1): number analyzed (Participants) | 20 | 0
  Total bacteria at baseline (S1) | 178500 [6210 to 2520000] |
  Total bacteria after root canal Preparation (S2): number analyzed (Participants) | 20 | 0
  Total bacteria after root canal Preparation (S2) | 7580 [0 to 835000] |
  Total bacteria after adjunctive procedures (S3): number analyzed (Participants) | 20 | 0
  Total bacteria after adjunctive procedures (S3) | 3815 [0 to 184000] |
  Total bacteria after intracanal medication (S4): number analyzed (Participants) | 20 | 0
  Total bacteria after intracanal medication (S4) | 15550 [0 to 209000] |
  Total bacteria after 2nd-visit preparation (S5): number analyzed (Participants) | 20 | 0
  Total bacteria after 2nd-visit preparation (S5) | 0 [0 to 96200] |
  Bacteroidaceae sp. 272 at S1: number analyzed (Participants) | 0 | 20
  Bacteroidaceae sp. 272 at S1 |  | 0 [0 to 320000]
  Bacteroidaceae sp. 272 at S2: number analyzed (Participants) | 0 | 20
  Bacteroidaceae sp. 272 at S2 |  | 0 [0 to 12300]
  Cutibacterium acnes at S1: number analyzed (Participants) | 0 | 20
  Cutibacterium acnes at S1 |  | 0 [0 to 17600]
  Cutibacterium acnes at S2: number analyzed (Participants) | 0 | 20
  Cutibacterium acnes at S2 |  | 0 [0 to 41400]
  Selenomonas spp. at S1: number analyzed (Participants) | 0 | 20
  Selenomonas spp. at S1 |  | 4090 [0 to 347000]
  Selenomonas spp. at S2: number analyzed (Participants) | 0 | 20
  Selenomonas spp. at S2 |  | 0 [0 to 3980]
  Enterococcus faecalis at S1: number analyzed (Participants) | 0 | 20
  Enterococcus faecalis at S1 |  | 0 [0 to 125000]
  Enterococcus faecalis at S2: number analyzed (Participants) | 0 | 20
  Enterococcus faecalis at S2 |  | 0 [0 to 0]

3. Secondary Outcome: Bacterial Community Diversity
Description: Composition of the active microbiome by Next Generation Sequencing (NGS) analysis of the root canal samples.
Time Frame: After 14 day treatment period
Population: Root canal samples from 10 patients were included in the sequencing analysis.
Measure: Number; unit: relative abundance of phyla (percentage)
Groups:
- Bacterial Composition at Baseline: Microbiome analysis in initial root canal samples by Next Generation Sequencing (NGS) based on RNA (cDNA).
- Bacterial Composition After Root Canal Preparation: Microbiome analysis in post-instrumentation samples by Next Generation Sequencing (NGS) based on RNA (cDNA).
- Bacterial Composition After Intracanal Medication: Microbiome analysis in post-medication samples by Next Generation Sequencing (NGS) based on RNA (cDNA).
Arm/Group | Bacterial Composition at Baseline | Bacterial Composition After Root Canal Preparation | Bacterial Composition After Intracanal Medication
Number analyzed (Participants) | 10 | 10 | 10
relative abundance of phyla (percentage)
  Firmicutes | 39.7 | 39.8 | 39.8
  Bacteroidetes | 39 | 39.1 | 38.6
  Proteobacteria | 15.8 | 15.7 | 16
  Actinobacteria | 1.4 | 1.4 | 1.6
  Spirochaetes | 0.7 | 0.7 | 0.6

4. Other Pre Specified Outcome: Endodontic Success
Description: Absence of clinical signs/ symptoms and reduction/ absence of apical radiolucency in radiologic examination
Time Frame: 1 year after endodontic treatment
Population: A subset of 30 patients had both intra-oral radiograph and cone beam computed tomography (CBCT) scans for analysis of the treatment outcome. After 1 year, 8 patients were lost during the follow-up period and 22 patients were analysed.
Measure: Count of Participants; unit: Participants
Groups:
- Root Canal Preparation and Medication: The success rate of the endodontic treatment after 1 follow-up period assessed by intraoral radiograph and cone beam computed tomography (CBCT) analyses.The number (%) of patients with absence/ reduction of periapical lesion are reported.
Arm/Group | Root Canal Preparation and Medication
Number analyzed (Participants) | 22
Participants | 19

ADVERSE EVENTS:
Time Frame: 0
Description: Adverse Events were not monitored/assessed because the endodontic treatment does not cause mortality or serious adverse events.
Groups:
- Root Canal Preparation and Medication: First endodontic treatment session includes the root canal preparation with Reciproc System and NaOCl 2.5%, followed by final irrigation protocol using activation techniques: XP Endo-Finisher and ultrasonic activation. The second endodontic treatment includes the intracanal medication with calcium hydroxide paste. Root canal samples from 20 patients were used to the analysis of total bacteria, Bacteroidaceae sp. HOT-272 and Cutibacterium acnes), while root canal samples from 25 patients were used for the analysis of total bacteria, Selenomonas spp. and Enterococcus faecalis
Arm/Group | Root Canal Preparation and Medication
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03537664/Prot_SAP_000.pdf